CLINICAL TRIAL: NCT03640468
Title: Lidocaine as an Adjuvant for Ketamine in Induction of Anesthesia in Septic Shock Patients: a Randomized Controlled Trial
Brief Title: Lidocaine as an Adjuvant for Ketamine in Induction of Anesthesia in Septic Shock Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor of anesthesia and critical care, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-128-2018
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Septic Shock; Anesthesia
MeSH Terms: conditions — Shock, Septic | interventions — Ketamine; Lidocaine; Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine group (Active Comparator): This group will receive induction of anesthesia using ketamie full dose 1 mg/kg, midazolam 0.05 mg/Kg, and normal saline 10 mL.
  Interventions: Drug: Ketamine full dose; Drug: Midazolam; Drug: Normal saline
- Lidocaine-ketamine group (Experimental): This group will receive induction of anesthesia using Ketamie half dose 0.5 mg/kg, midazolam 0.05 mg/Kg, and lidocaine 1 mg/Kg.
  Interventions: Drug: Ketamine half dose; Drug: Lidocaine; Drug: Midazolam

INTERVENTIONS:
Drug: Ketamine full dose — This group will receive induction of anesthesia using Ketamine 1 mg/Kg
  Other Names: Ketamine hydrochloride
  Arms: Ketamine group
Drug: Ketamine half dose — This group will receive induction of anesthesia using Ketamine 0.5 mg/Kg
  Other Names: Ketamine Hydrochloride
  Arms: Lidocaine-ketamine group
Drug: Lidocaine — This group will receive lidocaince 1 mg/Kg
  Other Names: Lidocaine Hydrochloride
  Arms: Lidocaine-ketamine group
Drug: Midazolam — This group will receive midazolam 0.05 mg/Kg
  Other Names: Dormicum
Drug: Normal saline — This group will receive normal saline 10 mL
  Arms: Ketamine group

SUMMARY:
The aim of the work is to investigate the effect of using lidocaine in combination with low dose ketamine in induction of anesthesia for septic shock patients compared to normal dose of ketamine.

DETAILED DESCRIPTION:
Most of the drugs used for induction of anesthesia negatively impact patient hemodynamics. Thus, induction of anesthesia in shocked patients might result in deleterious hypotension. Patients with severe sepsis and septic shock frequently need surgical interventions. The best protocol for induction of anesthesia in septic shock patients is lacking.

Ketamine is an agent used for induction of anesthesia with known positive cardiovascular effects. However, these positive effects were reported in individuals with intact sympathetic nervous system. Invitro studies showed that ketamine direct action on the cardiac muscles is negative. Thus, it had been recommended that ketamine should be used with caution in hemodynamically vulnerable patients till further randomized controlled trials are present.

Lidocaine is a drug with multiple local and systemic uses. Having local anesthetic properties, lidocaine was proposed to have an anesthetic sparing effect. Lidocaine was previously reported to enhance the hypnotic effect of thiopentone, propofol, and midazolam during induction of anesthesia. Lidocaine showed a sparing effect for volatile as well as intravenous requirements for maintenance of anesthesia; thus, we hypothesize that its use as an adjuvant during induction of anesthesia in septic shock patient could provide a sparing effect for ketamine and minimize its negative circulatory sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged above 18 years
* With septic shock
* Scheduled for general anesthesia

Exclusion Criteria:

* Patients under 18 years
* Burn patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-12-20 (Estimated); Primary Completion 2019-06-15 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure | 10 minutes after induction of general anesthesia
  Mean arterial pressure measured in mmHg

SECONDARY OUTCOMES:
Heart rate | 10 minutes after induction of general anesthesia
  number of heart beats per minutes
Cardiac output | 10 minutes after induction of general anesthesia
  volume of blood pumped by the heart in one minute measured in liters per minute
The number of patients who suffer from decreased mean arterial pressure by 20% from the baseline reading after induction of anesthesia | 10 minutes after induction of general anesthesia
Norepinephrine consumption | 10 minutes after induction of general anesthesia
  The total dose of norepinephrine measured in micrograms

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, Professor, Principal Investigator — Assistant professor of anesthesia
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No